CLINICAL TRIAL: NCT02720731
Title: Care-related Pain and Discomfort in Children and Adults With Motor Disorder in Medical Establishments
Brief Title: Care-related Pain and Discomfort in People With Motor Disorder
Acronym: DIS-HANDI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Brest (Other)
Collaborators: Fondation de France (Other); Fondation Motrice (Other); Fondation Apicil (Other)
Responsible Party: Sponsor
Other Study IDs: DIS-HANDI (RB 14.188)
Record Dates: First submitted 2016-03-10; First posted 2016-03-28 (Estimated); Last update posted 2016-07-12 (Estimated); Status verified 2016-07

CONDITIONS: Motor Disorders; Pain
MeSH Terms: conditions — Motor Disorders; Pain

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- children: aged from 1 to 18 years with motor disorder
- adults: aged from 18 to 80 years with motor disorder

SUMMARY:
The combination of motor disabilities, chronic pain, cognitive disabilities limiting the possibilities of communications and repeated potentially painful rehabilitation, exposes patients with motor disabilities to a high risk of induced pain in the specialized establishments. Induced pain is difficult to detect and is therefore little assessed and treated. Currently, little is known about the prevalence and conditions of occurrence of such induced pain as the clinical characteristics of patients (children, adults, severity of disability), the types of care and the nature of the institutional admission (medical or medico-social). Secondary objectives are to identify risk factors related to the induced pain and patient characteristics, as well as to create an easy-to-use weekly continuous pain assessment tool in a routine clinical set-up.

All daily life procedures or treatment carried out in children and adults with motor disability are collected for 5 days and 1 night. Collected data are clinical and demographic characteristics of patients, the intensity of the pain assessed by the care professional (FLACC-r) or the patient himself (VAS).

Clinically, the uncomfortable and painful procedures and risk factors for pain identified by this study will help the development of targeted preventive measures within institutions. Meanwhile, the study should sensitize Breton teams involved with regards to the induced pain, leading them to observe the behavior of patients, to admit any pain related to an act of daily life, and to ask for the medical profession to anticipate the painful experience.

ELIGIBILITY:
Inclusion Criteria:

* motor disorder
* institutionalized

Exclusion Criteria:

* chronical pain

Ages: 1 Year to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: children and adults with motor disorders admitted in medical institutions
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2016-04; Primary Completion 2017-11 (Estimated); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
Pain related to care-activities assessed with the Face, Legs, Activity, Cry, Consolability (FLACC-r) scale | 5 days

SECONDARY OUTCOMES:
Pain related to care-activities assessed with the Visual Analog Scale (VAS). | 5 days

CONTACTS AND LOCATIONS:
Overall Officials: sylvain BROCHARD, Study Director — Univesrity Hospital of Brest
Locations (10):
- France (10):
  - Centre Creac'h Ar Roual, Dirinon
  - IME section polyhandicapes Kerlaouen, Guipavas
  - SEAPH-IME Kerveguen, Plabennec
  - IEM Plerin, Plérin
  - IEM Ar Men, Ploemeur
  - Centre de Rééducation fonctionnelle de Kerpape, Ploemeur
  - CHRU de Rennes, Rennes
  - Fondation Ildys site de Perhardy, Roscoff
  - Centre Rééducation Trestel, Trévou-Tréguignec
  - EEAP Maison de L'estran, Trévou-Tréguignec